CLINICAL TRIAL: NCT02077075
Title: The Effectiveness of the MyHealthCheckup Wellness Program Among Canadian Forces Military Personnel
Brief Title: MyHealthCheckup Wellness Program Among Canadian Forces Military Personnel
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Steven Grover, MD, Director, McGill Comprehensive Health Improvement Program, McGill University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHIP13001
Record Dates: First submitted 2014-02-27; First posted 2014-03-04 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Overweight
Keywords: weight loss; healthy weight; overweight; body mass index greater that 25 kg/m2
MeSH Terms: conditions — Overweight; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Web-based weight loss program (Active Comparator): Subjects will have access to a web-based weight loss program for an 8-week period.
  Interventions: Behavioral: Web-based weight loss program
- On-line health coaching in addition to web-based program (Experimental): Subjects will have access to the web-based wellness program and will also receive weekly personalized health coaching emails.
  Interventions: Behavioral: Web-based weight loss program; Behavioral: On-line health coaching

INTERVENTIONS:
Behavioral: Web-based weight loss program — A 4-week web-based wellness program.
Behavioral: On-line health coaching — A 4-week web-based wellness program with weekly personalized on-line health coaching.
  Arms: On-line health coaching in addition to web-based program

SUMMARY:
This research is collecting data to determine the benefits of a web-based wellness program designed to improve the health and well-being of individuals in the workplace. Participants will be invited to participate in a web-based Healthy Weight Program. The program is designed to optimize health and wellbeing by promoting physical activity and healthy eating.

ELIGIBILITY:
Inclusion Criteria:

* A military member of the Canadian Forces Base in Halifax

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2014-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change in Body weight | 4 weeks
  Body weight

SECONDARY OUTCOMES:
Change in Waist circumference | 4 weeks
  Waist circumference measured at the umbilicus

CONTACTS AND LOCATIONS:
Overall Officials: Steven Grover, MD, Principal Investigator — McGill University
Locations (1):
- Canadian Forces Base Halifax, Halifax, Nova Scotia, Canada